CLINICAL TRIAL: NCT04288986
Title: The Impact of Group Based Activity Programmes on Children Who Have Autism and Their Families in Staffordshire
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Midlands Psychology CIC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MP/KA-3
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum condition; Autism; Sport; Wellbeing; Self-image
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The study will use a pretest-posttest quasi experimental design. Participants will complete a serious of questionnaires prior to participating in an 8 week activity programme and again after completing the programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Keep Achieving (KA) group (Experimental): Participants in the experimental group will take part in a 8-week group based activity programme. The activity programme will consist of 1, 50 minute session each week for the duration of 8-weeks. The activity sessions will include semi-structured free play sessions, sport specific sessions facilitated by local sports teams and swimming sessions.
  Interventions: Behavioral: Keep Achieving

INTERVENTIONS:
Behavioral: Keep Achieving — The 8-week group based activity programme will consist of 8 sessions each lasting 50 minutes.
  Other Names: 8-week group based activity programme

SUMMARY:
Participation in structured activities and physical activity (PA) have been linked to several indicators of positive development such as self-esteem and psychological health as well as greater academic outcomes and lower school drop-out rates. Despite this, 77% of boys and 80% of girls aged 5-15 in the UK also fall below the national physical activity guidelines of 60 minutes of moderate to vigorous activity per day.

Children with Autism Spectrum Conditions (ASC) may be at particular risk for inactivity as they are more likely to experience barriers to participation in these types of activities and motor skills impairments, common in people with ASC, can further limit participation in PA. Studies that have attempted to increase PA in young people with autism have shown reduction in problem behaviours such as inattention and aggression and increase in positive behaviours such as sleep, improvements in quality of life, academic performance and physical competence, and reductions in stress.

The primary research aim is to investigate whether participation in a 8-week group based activity programme affects social skills and problem behaviours in CYP with ASC.

DETAILED DESCRIPTION:
Participation in structured activities and physical activity (PA) have been linked to several indicators of positive development such as self-esteem and psychological health as well as greater academic outcomes and lower school drop-out rates. Despite this, 77% of boys and 80% of girls aged 5-15 in the UK also fall below the national physical activity guidelines of 60 minutes of moderate to vigorous activity per day.

Children with Autism Spectrum Conditions (ASC) may be at particular risk for inactivity. This group are more likely to experience barriers to participation in these types of activities and motor skills impairments, common in people with ASC, can further limit participation and enjoyment in PA and structured activities such as sports clubs and swimming lessons. Studies have shown that even at a young age children with ASC are less active than non-ASC children, and this physical activity gap gets wider as children get older.

Studies that have attempted to increase PA in young people with autism have shown reduction in problem behaviours such as inattention and aggression and increase in positive behaviours such as sleep, improvements in quality of life, academic performance and physical competence, and reductions in stress. However, many of these studies only worked with children 1:1 and therefore little is known about group-based activity intervention in young people with ASCs which could provide people with ASC opportunities to be physically active and as well as opportunities to socialise with others.

Parental modelling has been shown to be a predictor of children's PA behaviours with a positive correlation between adult and child PA levels. Given the influential role parents play on children's PA behaviours, parental involvement could be used as a function to increase PA in children with ASC.

It is not only young people with ASC who may struggle to access or fail to participate in sufficient PA but adults of the so called 'normal population'. In the UK, 34% of men and 42% of women do not meet the UK physical activity guidelines of 150 minutes of moderate activity per week. PA and civic participation may be particularly beneficial to parents of children with ASC as parents of children with developmental disorders have been shown to report lower quality of life, more depression, higher levels of stress anxiety, and greater pessimism about the future than parents of typically developing children. As a result, parents with children who have ASC may experience lower sense of connectedness to the social world.

Aims

To investigate whether participation in an 8-week group based activity programme affects social skills and problem behaviours in children and young people (CYP) with ASC.

Secondary aims

To investigate the effects of a weekly group based activity programme on parental wellbeing and social connectedness.

To investigate the effects of a weekly group based activity programme on CYP self-image.

To investigate parental goals for participating in a group based activity programme and evaluate progress toward these goals at the end of the programme.

To investigate session enjoyment levels from activities in the 8-week programme via a feedback form.

Hypotheses

There will be a difference in social skills and problem behaviours scores for CYP pre and post intervention.

There will be a difference in parental wellbeing and social connectedness scores for parents pre and post intervention.

There will be a difference in self-image scores for CYP pre and post intervention.

Method

Participants

The sample will consist of 20 CYP with an ASC and 20 parents/carers of CYP with an ASC. All participants will take place in an 8-week group based activity programme.

Principle inclusion criteria include; children with a working or full ASC diagnosis aged between 5-15 years, self-declared physically fit to participate in activities. Siblings and additional adults will also be invited to participate in the programme in order to support their sibling with ASC and to make attendance easier for parents who would otherwise struggle with childcare if they were not able to participate in the programme as a family. However, data will not be collected from this group. Participants will be recruited through advertisements on social media and at local autism support groups.

Design

The study will use a pretest-posttest quasi experimental design. Participants will complete a serious of questionnaires prior to participating in an 8 week activity programme and again after completing the programme.

The 8-week group based activity programme will consist of 8 sessions each lasting 50 minutes. The sessions in the programme will be different each week. A number of sessions will be semi-structured free play sessions which will be supervised by qualified staff from Midlands Psychology CIC; 2 assistant psychologists and a project manager. All staff will have enhanced DBS checks and over a years' experience running these kinds of activity sessions with families. Risk assessments will be completed prior to each session.

Semi-structured free play sessions will be consist of a range of activities which parents and CYP can participate in together (frisbee, hockey, soft play, football, obstacle courses, glow in the dark activities).

Several sessions will be hosted by local sports clubs such as football, rugby and handball. When sports clubs host session they will be instructed to break their sport down into a series fun 'drills' for families to participate in such as passing skills, dribbling, shooting, ending with a small game.

There will be a swimming session taking place in the swimming pool of a local leisure centre. For this session parents and CYP will be supervised in the swimming pool by trained lifeguards and staff members from Midlands Psychology CIC will not be in the swimming pool.

The final session in the programme will be a novel activity such as a climbing session at a 'clip and climb' centre to celebrate participation in the programme. This session will be run by the centres' own staff, who have experience running these sessions and require families to participate in a safety briefing and demonstration prior to climbing.

Participants can choose to participate in a group based activity programme running in either Stafford, Burton, Cannock or Tamworth.

Procedure

Participants will be recruited via online advertisements. These advertisements will target families living within the Staffordshire area. The advertisements will inform prospective participants of the 8-week group based programme and ask all interested to contact the research team for further information.

Participants will be sent (via email or post if requested) a parent and child information sheet detailing what the study entails and the consent and assent forms to be completed for all those taking part in the research. Participants will be informed that they can drop out of the study at any time and ask for their data to be withdrawn. Participants will also have the opportunity to contact the researchers and have any queries addressed.

Prior to the start of the activity programme, all participants will have the oppourtunity to complete the following measures with the researchers or have them sent in the post; the Social Skills Improvement System -Parent (SSIS), Social Skills Improvement System -Student (SSIS), Social Connectedness Scale - Revised (SCS-R), Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS), the Self Image Profile (SIP) and goal based outcomes (GBO). If participants have these sent via post, they will be asked to return all of these prior to the start of the 8-week activity programme. Once the 8-week activity programme has ended, participants will again be asked to complete the SSIS, SCS-R, SWEMWBS, SIP and GBOs. Participants will be thanked for their participation in the research.

For children under the age of 8 years, only their parents' data will be collected as the questionnaires require a minimum age of 8.

Measures

Social Skills Improvement System Rating Scales. For both adults and CYP (CYP over the age of 8)

The Social Skills Improvement System (SSIS) evaluates social skills and problem behaviours. There are two separate questionnaires: one for parents/guardians and one for CYP. Parents/guardians report on the frequency their children exhibit social skills and problem behaviours on a 4-point scale: never, seldom, often, and almost always.

Social Connectedness Scale Revised

For adults only

Social Connectedness is considered is an attribute of the self, reflecting interpersonal thoughts and closeness to the social world. The scale is comprised of 10 negatively worked and 10 positively worded items such as "I feel comfortable in the presence of strangers" and "I feel myself as an outsider". Participants rate the degree to which they agree or disagree on a scale from 1-6 (1= strongly disagree, 6 strongly agree).

The Short Warwick-Edinburgh Mental Wellbeing Scales (SWEMWBS)

For adults only

The Short version of the Warwick-Edinburgh Mental Wellbeing Scales measures positive aspects of mental health in the prior 2 weeks such as "i've been feeling useful" or "i've been feeling relaxed". The scale comprises 7 positively phrased items responded on a 5-point Likert-type scale from 'None of the time' to 'All of the time'.

Self Image Profile

For children only

This SIP invites respondents to give two ratings of how they consider themselves to be; and how they would like to be across 25 items. Participants rate each item from 0 (Not At All) to 6 (Very Much). The SIP comprises 12 items of a positive nature i.e. 'Intelligent' and 12 of a negative tone 'mess about'. Once completed a self image score (summation of the first rating) and self esteem score (operationally defined as the discrepancy between the two ratings) can be obtained.

Goal Based Outcomes (GBOs)

For adults only

Parents will be asked to state 3 goals that they wish to achieve from participating in the 8-week programme. Prior to the start of the intervention, parents will be asked to rate where they feel they are now in relation to achieving a specified goal on a scale of 0-10, 0 being 'goal not at all met' and 10 being 'goal reached'. At the end of the intervention, parents will be asked to again rate where they feel they are now in relation to achieving a specified goal on the same rating scale.

Proposed data analysis SSIS (Social Skills and Problem Behaviours) A paired-samples t-test will be used to compare the pre-test and post-test scores for social skills and problem behaviours on the parental SSIS.

A paired-samples t-test will be used to compare the pre-test and post-test scores for social skills and problem behaviours on the student SSIS.

SIP (Self-image)

A paired-samples t-test will be used to compare the pre-test and post-test scores for self-image for children with ASC.

SWEMWBS (Wellbeing)

A paired-samples t-test will be used to compare the pre-test and post-test scores for parental mental wellbeing.

SCS-R (Social Connectedness) A paired-samples t-test will be used to compare the pre-test and post-test scores for parents' feelings of social connectedness.

GBO's (Goal Based Outcomes) The GBO ratings from pre and post-intervention for the experimental group will be compared to investigate to what extent parents felt their goals for participation were reached.

Enjoyment The enjoyment ratings will be correlated with session attendance figures to see whether attendance in the 8-week programme was associated with enjoyment of the sessions.

ELIGIBILITY:
Inclusion Criteria:

* A child or young person with a working or full diagnosis of an Autism spectrum condition (ASC). Parents/carers will be asked to provide proof in the form of a letter that their child has an ASC.

The child with an ASC must be between the ages of 5-15 years. All participants must confirm they are physically fit to participate in this research as some activities involve moderate to vigorous physical activity.

All children with an ASC who are receiving alternative support are required to declare this prior to participation and specify the type of support received.

Exclusion Criteria:

* Children/young people without a full or working ASC diagnosis Children with a full or working diagnosis of ASC not between the ages of 5-15 years People who are not deemed physically fit to participate in the activity programme by their own self-assessment.

Current or recent participation in another clinical trial/study/scientific experiment

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Social Skills Improvement System Rating Scales - Parent (SSIS; Gresham & Elliott (2007). | 14 weeks
  The Social Skills Improvement System (SSIS) evaluates social skills and problem behaviours. Parents/guardians report on the frequency their children exhibit social skills and problem behaviours on a 4-point scale: never, seldom, often, and almost always. Social skills are evaluated in the following domains: communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. Problem behaviours assessed include: externalizing, bullying, hyperactivity/inattention, internalising, and "autism spectrum".
Social Skills Improvement System Rating Scales - Child (SSIS; Gresham & Elliott (2007). | 14 weeks
  The Social Skills Improvement System (SSIS) evaluates social skills and problem behaviours. Young people (8-18) indicate if a variety of different statements about problem behaviours or social skills are true of them on a 4-point scale: not true, a little true, a lot true, and very true. Social skills are evaluated in the following domains: communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. Problem behaviours assessed include: externalizing, bullying, hyperactivity/inattention, internalising, and "autism spectrum".

SECONDARY OUTCOMES:
Social Connectedness Scale Revised (SCS-R; Lee, Draper & Lee 2001) | 14 weeks
  Social Connectedness is considered is an attribute of the self, reflecting interpersonal thoughts and closeness to the social world. The scale is comprised of 10 negatively worked and 10 positively worded items such as "I feel comfortable in the presence of strangers" and "I feel myself as an outsider". Participants rate the degree to which they agree or disagree on a scale from 1-6 (1= strongly disagree, 6 strongly agree).
Self Image Profile (SIP; Butler) | 14 weeks
  This SIP invites respondents to give two ratings of how they consider themselves to be; and how they would like to be across 25 items. Participants rate each item from 0 (Not At All) to 6 (Very Much). The SIP comprises 12 items of a positive nature i.e. 'Intelligent' and 12 of a negative tone 'mess about'. Once completed a self image score (summation of the first rating) and self esteem score (operationally defined as the discrepancy between the two ratings) can be obtained.
The Short Warwick-Edinburgh Mental Wellbeing Scales (SWEMWBS; Stewart-Brown et al., 2009) | 14 weeks
  The Short version of the Warwick-Edinburgh Mental Wellbeing Scales measures positive aspects of mental health in the prior 2 weeks such as "i've been feeling useful" or "i've been feeling relaxed". The scale comprises 7 positively phrased items responded on a 5-point Likert-type scale from 'None of the time' to 'All of the time'.
Goal Based Outcomes (GBOs) | 14 weeks
  Parents will be asked to state 3 goals that they wish to achieve from participating in the 8-week programme. Prior to the start of the intervention, parents will be asked to rate where they feel they are now in relation to achieving a specified goal on a scale of 0-10, 0 being 'goal not at all met' and 10 being 'goal reached'. At the end of the intervention, parents will be asked to again rate where they feel they are now in relation to achieving a specified goal on the same rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: James Smolinski, MSc, Principal Investigator — james.smolinski@midlandspsychology.co.uk
Locations (1):
- The Hates, Stafford, Staffs, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eccles, J. S., & Barber, B. L. (1999). Student council, volunteering, basketball, or marching band what kind of extracurricular involvement matters? Journal of adolescent research, 14(1), 10-43.
- [Background] Hastings RP, Kovshoff H, Ward NJ, degli Espinosa F, Brown T, Remington B. Systems analysis of stress and positive perceptions in mothers and fathers of pre-school children with autism. J Autism Dev Disord. 2005 Oct;35(5):635-44. doi: 10.1007/s10803-005-0007-8. PMID 16177837
- [Background] Kohl HW 3rd, Hobbs KE. Development of physical activity behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):549-54. PMID 12224661
- [Background] Lang, R., Koegel, L. K., Ashbaugh, K. et al. (2010). Physical exercise and individuals with autism spectrum disorders: A systematic review. Research in Autism Spectrum Disorders, 4(4), 565-576.
- [Background] Lee, R. M., Draper, M., & Lee, S. (2001). Social connectedness, dysfunctional interpersonal behaviors, and psychological distress: Testing a mediator model. Journal of counseling psychology, 48(3), 310.
- [Background] Neff, K. D., & Faso, D. J. (2015). Self-compassion and well-being in parents of children with autism. Mindfulness, 6(4), 938-947.
- [Background] Memari, A. H., Kordi, R., Ziaee, V. (2012). Weight status in Iranian children with autism spectrum disorders: Investigation of underweight, overweight and obesity. Research in Autism Spectrum Disorders, 6(1), 234-239.
- [Background] Public Health England (2016). Health matters: getting every adult active every day. [online] Available at: https://www.gov.uk/government/publications/health-matters-getting-every-adult-active-every-day/health-matters-getting-every-adult-active-every-day [Accessed 20 Aug. 2019].
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Trost SG, Kerr LM, Ward DS, Pate RR. Physical activity and determinants of physical activity in obese and non-obese children. Int J Obes Relat Metab Disord. 2001 Jun;25(6):822-9. doi: 10.1038/sj.ijo.0801621. PMID 11439296
- [Result] Butler R.J. (2001) The self-image profile for children (SIP-C) and adolescents (SIP-A). Manual. London, The Psychological Corporation